CLINICAL TRIAL: NCT06479421
Title: A Clinical Study for Developing AI-based Clustering Model for Personalized Medicine in Acute Respiratory Failure: Single Center, Prospective Cohort Study
Brief Title: A Clinical Study for Developing Artificial Intelligence(AI)-Based Clustering Model for Personalized Medicine in Acute Respiratory Failure
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: Ministry of Science and ICT, Republic of Korea (Other Government)
Responsible Party: Principal Investigator, Ryoung-Eun Ko, Clinical assistant professor, Samsung Medical Center
Other Study IDs: 2023-08-003
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Acute Respiratory Failure
Keywords: phenotyping; clustering analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. Blood sample collection
     : Within 24 hours after admission to the intensive care unit, and 2 to 5 days after admission to the intensive care unit, 18 ml of blood is collected in an ethylenediaminetetraacetic acid(EDTA) tube once (a total of 2 times, 36 ml) to analyze the following.
     * Interleukin(IL)-6, IL-8, tumor necrosis factor receptor-1 levels, etc. will be checked.
     * If the planned sample collection time has passed after admission to the intensive care unit or if blood sample collection is difficult due to quarantine, etc., this can be omitted.
  2. Broncho-Alveolar Lavage(BAL) fluid sample collection
     * Only for those subjects who undergo BAL during the treatment process, 5ml of BAL fluid will be collected and analyzed for the following.
       * IL-1β, IL-6, IL-8, Kerbs von Lungren-6, Plasminogen activator inhibitor-1, etc. will be checked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute Respiratory Failure group: Among patients admitted to the internal medicine intensive care unit at Samsung Seoul Hospital, if all of the following conditions are met:
  1. Age 18 or older
  2. Patients who require treatment with high flow nasal cannula (HFNC), non-invasive ventilation (NIV (BIPAP or CPAP)), or mechanical ventilation (MV) due to acute respiratory failure.
- Control group: For comparative analysis, among patients admitted to the internal medicine intensive care unit at Samsung Seoul Hospital who meet all of the following conditions, they are registered as a control group with the consent of the subjects and undergo the same research procedure.
  1. Age 18 or older
  2. Patients who do not require high flow nasal cannula (HFNC), non-invasive ventilation (NIV (BIPAP or CPAP)), or mechanical ventilation (MV) treatment

SUMMARY:
We will prospectively collect clinical information to develop a clustering analysis model and confirm phenotype for patients with acute respiratory failure who admit to the intensive care unit and require oxygen supply beyond a high flow nasal cannula, and a control group without acute respiratory failure. and clinical characteristics and prognosis will be compared.

ELIGIBILITY:
# Inclusion Criteria:

- Acute Respiratory Failure group

Among patients admitted to the internal medicine intensive care unit at Samsung Seoul Hospital, if all of the following conditions are met:

1) Age 18 or older 2) Patients who require treatment with high flow nasal cannula (HFNC), non-invasive ventilation (NIV (BIPAP or CPAP)), or mechanical ventilation (MV) due to acute respiratory failure.

- control group For comparative analysis, among patients admitted to the internal medicine intensive care unit at Samsung Seoul Hospital who meet all of the following conditions, they are registered as a control group with the consent of the subjects and undergo the same research procedure.

1. Age 18 or older
2. Patients who do not require high flow nasal cannula (HFNC), non-invasive ventilation (NIV (BIPAP or CPAP)), or mechanical ventilation (MV) treatment

   * Exclusion Criteria:

If any of the following criteria applies, you will not be permitted to participate in this clinical trial.

1. Patients 48 hours after oxygen treatment (HFNC, NIV (BIPAP or CPAP), MV)
2. Patients transferred from another hospital
3. Patients with limitations in treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients with acute respiratory failure admitted to the internal medicine intensive care unit of Samsung Seoul Hospital 1) Age 18 or older 2) Patients who require treatment with high flow nasal cannula (HFNC), non-invasive ventilation (NIV (BIPAP or CPAP)), or mechanical ventilation (MV) due to acute respiratory failure.
  2. The following patients (control group) admitted to the internal medicine intensive care unit of Samsung Seoul Hospital 1) Age 18 or older 2) Patients who do not require high flow nasal cannula (HFNC), non-invasive ventilation (NIV (BIPAP or CPAP)), or mechanical ventilation (MV) treatment
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Hospital Mortality | From date of admission until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 1 year
  clinical outcomes - Hospital Mortality

SECONDARY OUTCOMES:
ICU Mortality | From date of ICU admission until the date of ICU discharge or date of death from any cause, whichever came first, assessed up to 6 months
  clinical outcomes - ICU Mortality
Hospital length of stay | From date of hospital admission until the date of hospital discharge, assessed up to 1 years
  clinical outcomes - Hospital length of stay
ICU length of stay | From date of ICU admission until the date of ICU discharge, assessed up to 6 months
  clinical outcomes - ICU length of stay

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Gangnam, South Korea

IPD SHARING:
Plan to Share IPD: Undecided